CLINICAL TRIAL: NCT05103215
Title: The Analgesic Effect of Intravenous Lidocaine Infusion in Combination of Analgesia Nociception Index Monitoring in Spine Surgery.
Brief Title: Lidocaine Infusion With ANI Monitoring in Spine Surgery.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20210157
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Spine Surgery
Keywords: Lidocaine, enhanced recovery after surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine group (Experimental): Patients in the lidocaine group receive an intravenous injection of 1.5 mg/kg Lidocaine HCl 2% at induction of anesthesia and continuous infusion of 1.5 mg/kg/h (ideal body weight) through the maintenance period to one hour after operation.
  Interventions: Drug: Lidocaine HCl 2%
- control group (Placebo Comparator): Patients in control group receive the same volume of saline injection.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine HCl 2% — Intravenous injection of 1.5 mg/kg lidocaine at induction of anesthesia and continuous infusion of 1.5 mg/kg/h (ideal body weight) through the maintenance period to one hour after operation.
  Other Names: Xylocaine Injection 2%
  Arms: lidocaine group
Drug: Normal saline — Intravenous injection of 1.5 mg/kg normal saline at induction of anesthesia and continuous infusion of 1.5 mg/kg/h (ideal body weight) through the maintenance period to one hour after operation.
  Other Names: 0.9% Normal Saline (20mL)
  Arms: control group

SUMMARY:
To evaluate the analgesic effect of intraoperative continuous lidocaine infusion (1.5 mg/kg/h (ideal body weight)) in combination of analgesia nociception index and depth of anesthesia monitors guided anesthetics adjustment on enhanced recovery after surgery (ERAS) in patients undergoing elective lumbar spine surgery (≥2 sessions).

DETAILED DESCRIPTION:
The patients undergoing elective lumbar spine surgery (≥2 sessions) are randomly assigned and divided patients into two groups according to the allocation sequence table (corresponding to 1:1 randomization) generated by the computer. Patients in the lidocaine group receive an intravenous injection of 1.5 mg/kg lidocaine at induction of anesthesia and continuous infusion of 1.5 mg/kg/h (ideal body weight) through the maintenance period to one hour after operation. Patients in control group receive the same volume of saline injection. During the operation, the dose of anesthetic drugs (propofol, remifentanil and rocuronium) are adjusted to maintain the mean arterial pressure and heartbeat fluctuations within 20% of the baseline value, Entropy (or BIS) value at 40-60, and ANI at 50-70 in both groups. The pain score (numerical rating scale), cumulative amount of opioids used after the operation within 3 days, and the quality of recovery on the third day after the operation are recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Twenty to eighty-year-old
2. ASA class I-III patients undergoing
3. Elective lumbar spine surgery under general anesthesia

Exclusion Criteria:

1. Unable to understand the Numerical Rating Scale (NRS)
2. Severe mental disorder
3. Poor liver function
4. Pregnant or lactating women
5. Morbidly obese
6. History of epilepsy or allergy to any of the drugs used in this study
7. Current use of opioids
8. Baseline heart rate <50 beats/min
9. Arrhythmia history with cardiac rhythm device
10. Body weight <40 kg and >80kg

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
cumulative amount of opioids used | within 48 hours after operation
  cumulative amount of opioids used after the operation
the quality of recovery after the operation | on the third day after the operation
  Quality of recovery-15 score, QoR-15, 0-150, higher score means better outcome
pain score | within 72 hours after operation
  numerical rating scale, NRS, 0-10, higher score means worse outcome

SECONDARY OUTCOMES:
cumulative amount of opioids used | within 72 hours after operation
  cumulative amount of opioids used after the operation
cumulative amount of propofol used | during operation
  cumulative amount of propofol used
cumulative amount of remifentanil used | during operation
  cumulative amount of remifentanil used
cumulative amount of rocuronium used | during operation
  cumulative amount of rocuronium used

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Fu Wu, MD, Study Chair — Kaohsiung Medical University Hospital, Kaohsiung Medical University, Kaohsiung City, Taiwan (R.O.C.)
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No